CLINICAL TRIAL: NCT01940952
Title: Efficacy of Zydena (Udenafil) on Cognitive Function of Alzheimer's Disease Patients: A Randomized, Double Blind, Placebo-controlled Multicenter Study
Brief Title: Zydena on Cognitive Function of Alzheimer's Disease Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Duk Lyul Na, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-03-065; 2012-03-065 (Other: Samsung Medical Center)
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — udenafil; Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Zydena 50mg (Active Comparator): Zydena (Udenafil) 50mg + Donepezil 5mg or 10mg
  Interventions: Drug: Zydena (Udenafil) 50mg + Donepezil 5mg or 10mg
- Placebo (Placebo Comparator): Placebo + Donepezil 5mg or 10mg
  Interventions: Drug: Placebo + Donepezil 5mg or 10mg
- Zydena 100mg (Active Comparator): Zydena (Udenafil) 100mg + Donepezil 5mg or 10mg
  Interventions: Drug: Zydena (Udenafil) 100mg + Donepezil 5mg or 10mg

INTERVENTIONS:
Drug: Zydena (Udenafil) 50mg + Donepezil 5mg or 10mg
  Other Names: Zydena 50mg
  Arms: Zydena 50mg
Drug: Placebo + Donepezil 5mg or 10mg
  Other Names: Placebo
  Arms: Placebo
Drug: Zydena (Udenafil) 100mg + Donepezil 5mg or 10mg
  Other Names: Zydena 100mg
  Arms: Zydena 100mg

SUMMARY:
The purpose of this study is to determine whether Zydena (Udenafil) has positive effect on cognitive function in patients with Alzheimer's disease.

This study is a randomized, double blind, placebo-controlled multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent;
* Male or female subjects 50 to 90 years of age;
* Diagnosis of probable Alzheimer's disease according to National Institute of Neurological Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria;
* A Mini-Mental State Examination (MMSE) score of ≥10 and ≤26;
* Global Clinical Dementia Rating ≥ 0.5;
* Mild to moderate (not severe) white matter hyperintensities on brain MRI performed within three years from screening;
* Good enough hearing and visual function to complete neuropsychological tests
* Caregivers living with patients or spending 10 or more hours a week with patients;
* Stable dose of donepezil (5mg to 10mg) for at least 60 days;
* If patients have been on memantine, it should be washed out for at least 60 days;
* Medications including anxiolytics, antipsychotics, and hypnotics may be taken if the dose has been stable for at least two weeks

Exclusion Criteria:

* History of stroke within 6 months;
* Previous diagnosis of severe (more than 80%) intracranial artery stenosis;
* History of heart failure, ischemic heart disease (myocardial infarction, unstable angina, and stable angina), hypertrophic cardiomyopathy, and life-threatening arrhythmia;
* Previous history of coronary artery bypass graft surgery;
* Severe symptom of orthostatic hypotension (orthostatic syncope or presyncope), especially when patients take alpha-adrenergic blocker (Alfuzosin, Doxazosin, Naftopidil, Tamsulosin, Terazosin, Arotinolol, Carvedilol, Labetalol, Trazodone, typical and atypical antipsychotics);
* Uncontrolled diabetes mellitus;
* Proliferative diabetic retinopathy;
* Severe hypotension (blood pressure less than 90/50mmHg) or severe hypertension (blood pressure more than 170/100mmHg);
* Hepatic dysfunction (AST or ALT more than three times of upper normal limit) or renal dysfunction (serum creatinine more than 2.5mg/dL);
* Retinitis pigmentosa;
* Previous history of active peptic ulceration within one year before screening;
* Hematodyscrasia susceptible to priapism including sickle cell anemia, multiple myeloma, leukemia, and various bleeding disorders;
* History of drug abuse;
* Medication including nitrates/nitric oxide donor (ex: nitroglycerin, isosorbide mononitrate, isosorbide dinitrate, amyl nitrate/nitrite, and Sodium nitroprusside), androgen (ex: testosterone), anti-androgen, and anticoagulants;
* Current cancer chemotherapy;
* Usage of PDE5i (Zydena, Viagra®, Levitra®, or Cialis®) within two weeks before study start;
* History of hypersensitive reaction to PDE5i (Zydena, Viagra®, Levitra®, or Cialis®)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive function | from baseline to Week 12 and Week 24 after the administration of the medication
  measured by ADAS-cog

SECONDARY OUTCOMES:
Change in cognitive function | from baseline to Week 12 and Week 24
  Measured by MMSE, Clinical Dementia Rating Sum of Boxes, ADCS-ADL, COWAT, Digit Symbol Coding, Trail Making Test-E
Change in behavioral symptoms | from baseline to Week 12 and Week 24
  Measured by Neuropsychiatric Inventory
Change in brain function | from baseline to Week 12 and Week 24
  Measured by FDG-PET

CONTACTS AND LOCATIONS:
Locations (1):
- Samguns Medical Center, Seoul, South Korea